CLINICAL TRIAL: NCT02431637
Title: Blood Stage Challenge Study to Asses Mosquito Transmissibility in Participants Inoculated With Plasmodium Falciparum
Brief Title: Experimental Falciparum Transmission to Anopheles
Acronym: EFITA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Q-Pharm Pty Limited (Industry); Clinical Network Services (CNS) Pty Ltd (Industry); Sullivan Nicolaides Pathology (Industry); QIMR Berghofer Medical Research Institute (Other); Army Malaria Institute, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QP14C21
Record Dates: First submitted 2015-04-17; First posted 2015-05-01 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Malaria
Keywords: Induced blood stage malaria; Transmission; Standard membrane feeding assay
MeSH Terms: conditions — Malaria | interventions — piperaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Piperaquine Phosphate after infected blood malaria challenge (Experimental): Volunteers will receive a dose of 480 mg piperaquine phosphate (PQP) approx. 7 days after a challenge with P. falciparum infected red blood cells. The effects of PQP on gametocyte carriage (assessed by PCR) and infectivity to mosquitos after direct and indirect feeding on blood from volunteers will be assessed.
  Interventions: Biological: Administration of the malaria inoculum; Drug: Piperaquine Phosphate 480 mg

INTERVENTIONS:
Biological: Administration of the malaria inoculum — Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. The threshold for commencement of treatment will be when PCR quantification of all participants is ≥ 5,000 parasites/mL.
Drug: Piperaquine Phosphate 480 mg — When PCR quantification of all participants is ≥ 5,000 parasites/mL, participants will receive a single dose of 480 mg Piperaquine Phosphate

SUMMARY:
This is a single-centre, open-label study using P. falciparum-induced blood stage malaria (IBSM) infection to assess the infectivity of sexual life cycle stages of the malaria parasite (gametocytes) to mosquito vectors. Previous clinical studies have shown that treatment of participants with the antimalarial drug piperaquine, in addition to effectively clearing asexual (pathogenic) stages of the malaria life cycle, induces the production of gametocytes in the blood. The propensity of piperaquine to induce gametocytemia will be employed in this study to assess gametocyte infectivity to Anopheles mosquitoes. For this purpose, experimental mosquito feeding directly on participants and artificial membrane mosquito feeding will be performed. The study will be conducted in 3 cohorts (n=2 per cohort). Subsequent cohorts will not commence until at least after day 28 of the previous cohort and review by Safety Review Team. This interval will also allow cohorting of experimental infection of mosquitoes to optimise logistics and enable iterative improvements in the system if applicable.

DETAILED DESCRIPTION:
This is a single-centre, open-label study using P. falciparum-induced blood stage malaria (IBSM) infection to assess the infectivity of sexual life cycle stages of the malaria parasite (gametocytes) to mosquito vectors. Previous clinical studies have shown that treatment of participants with the antimalarial drug piperaquine, in addition to effectively clearing asexual (pathogenic) stages of the malaria life cycle, induces the production of gametocytes in the blood. The propensity of piperaquine to induce gametocytemia will be employed in this study to assess gametocyte infectivity to Anopheles mosquitoes. For this purpose, experimental mosquito feeding directly on participants and artificial membrane mosquito feeding will be performed. The study will be conducted in 3 cohorts (n=2 per cohort). Subsequent cohorts will not commence until at least after day 28 of the previous cohort and review by Safety Review Team. This interval will also allow cohorting of experimental infection of mosquitoes to optimise logistics and enable iterative improvements in the system if applicable.

Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. On an outpatient basis, participants will be monitored daily via phone call and then daily (AM) from day 4 (until PCR positive for presence of malaria parasites). Once PCR positive they will be monitored twice-daily morning (AM) and evening (PM) until treatment, for adverse events and the unexpected early onset of symptoms, signs or parasitological evidence of malaria. On the day designated for commencement of treatment, as determined by qPCR results (approximately day 6-8), participants will be admitted to the study unit and monitored. The threshold for commencement of treatment will be when PCR quantification of all participants is = 5,000 parasites/mL. If the PCR quantification of any participant is = 10,000 parasites/mL and is accompanied by a clinical symptom score >8 occurs in any participant before all participants have reached the treatment threshold (PCR quantification of = 5,000), then treatment of that participant will begin within a 24 h period. Participants will be followed up as inpatients for at least 48 hours to ensure tolerance of the treatment and clinical response, then if clinically well on an outpatient basis for safety and clearance of malaria parasites via PCR.

Following treatment with piperaquine, transmission studies will be undertaken when gametocytemia appears. Blood will be collected (AM) from each participant for membrane feeding assays with An. Stephensi. For membrane feeding studies, blood will be kept at 38C (to prevent premature exflagellation) for up to 35 minutes until dispensed into membrane feeders. For direct feeding studies, participants will be escorted to the quarantine insectary facility at QIMR Berghofer and will also be asked to allow vector mosquitoes to feed on the volar surface of their forearms or thighs for a period of 10 ± 5 minutes (direct feeding assay). The experimental infection of mosquitoes by direct feeding on participants will be performed up to 3 times, and by artificial (indirect) membrane feeding up to 10 times prior to curative antimalarial treatment at the End Of Study with Riamet® (artemether-lumefantrine) and primaquine (45 mg).

A repeat dose of piperaquine 960 mg may be administered on an outpatient basis if recrudescent asexual parasitemia occurs as defined by consecutively increasing parasite count over 1000 parasites/mL. Preemptive rescue treatment with Riamet® can commence whenever deemed necessary by the investigator. Participants can be administered the rescue Riamet® on site for initial dosing followed by monitoring, either in clinic, or by telephone for three days to ensure adherence to Riamet® therapy.

Participants will be treated with a single dose of primaquine (45 mg) as described in section 4.4.2 in this protocol concurrent with their Riamet® treatment to ensure clearance of any gametocytes present.

Adverse events will be monitored via telephone monitoring, within the clinical research unit, and on outpatient review after malaria challenge inoculation and anti-malarial study drugs administration. Blood samples for safety evaluation, malaria monitoring, and red blood cell antibodies will be drawn at screening and/or baseline and at nominated times after malaria challenge.

ELIGIBILITY:
Inclusion Criteria:

Demography:

* Adult (male and females) participants between 18 and 55 years of age, inclusive who do not live alone (from Day 0 until at least the end of the anti-malarial drug treatment) and be contactable and available for the duration of the trial (maximum of 6 weeks).
* Body weight, minimum 50.0 kg, body mass index between 18.0 and 32.0 kg/m

Health status:

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position:
* 90mmHg < systolic blood pressure (SBP) <140 mmHg,
* 50 mmHg < diastolic blood pressure (DBP) <90 mmHg,
* 40 bpm< heart rate (HR) <100 bpm.
* Normal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position, QTcF=450 ms average with absence of second or third degree atrioventricular block or abnormal T wave morphology.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants enrolled in this clinical investigation. More specifically for serum creatinine, hepatic transaminase enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the Participant has documented Gilbert syndrome) should not exceed the upper laboratory norm and haemoglobin must be equal or higher than the lower limit of the normal range, - - As the safety of Piperaquine on foetal development is unknown it is important that any participants involved in this study do not get pregnant or get their female partners pregnant.

Regulations:

- Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

Medical history and clinical status:

* Any history of malaria or participation to a previous malaria challenge study
* Must not have travelled to or lived (>2 weeks) in a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* Known severe reaction to mosquito bites other than local itching and redness
* Has evidence of increased cardiovascular disease risk (defined as >10%, 5 year risk) as determined by the method of Gaziano et al. (1). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, body mass index (BMI, kg/m) and reported diabetes status.
* History of splenectomy.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin-dependent and NIDDM diabetes (excluding glucose intolerance if E04 is met ), progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma
* Participants with history of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis including depression or receiving psychiatric drugs or who has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Frequent headaches and/or migraine, recurrent nausea, and/or vomiting (more than twice a month).
* Presence of acute infectious disease or fever (e.g., sub-lingual temperature = 38.5°C) within the five days prior to inoculation with malaria parasites.
* Evidence of acute illness within the four weeks before trial prior to screening that the Investigator deems may compromise subject safety.
* Significant intercurrent disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
* Participant has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhoea.
* Participation in any investigational product study within the 12 weeks preceding the study.
* Blood donation, any volume, within 1 month before inclusion or participation in any research study involving to be desired blood sampling (more than 450 mL/ unit of blood), or blood donation to Red Cross (or other) blood bank during the 8 weeks preceding the reference drug dose in the study.
* Participant unwilling to defer blood donations for 6 months.
* Medical requirement for intravenous immunoglobulin or blood transfusions.
* Participant who has ever received a blood transfusion.
* Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure =20 mmHg within 2-3 minutes when changing from supine to standing position.
* History or presence of alcohol abuse (alcohol consumption more than 40 g per day, 3 standard drinks per day) or drug habituation, or any prior intravenous usage of an illicit substance.
* Smoking more than 5 cigarettes or equivalent per day and unable to stop smoking for the duration of the study.
* Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (participants will
* be advised by phone not to consume any poppy seeds in this time period).

Interfering substance:

* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the
* elimination half-life (whichever is longer) of the medication,
* Any vaccination within the last 28 days.
* Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants. Any
* participant currently receiving or having previously received immunosuppressive therapy,
* including systemic steroids including adrenocorticotrophic hormone (ACTH) or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression such as 1mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids (budesonide 800 µg per day or fluticasone 750 µg).
* Any recent or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (chloroquine, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, hydroxychloroquine, etc.).

General conditions:

* Any participant who, in the judgment of the Investigator, is likely to be non compliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any participant in the exclusion period of a previous study according to applicable regulations.
* Any participant who lives alone (from Day 0 until at least the end of the anti-malarial drug treatment).
* Any participant who cannot be contacted in case of emergency for the duration of the trial and up to 2 weeks following end of study visit.
* Any participant who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Any participant without a good peripheral venous access.

Biological status:

* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human-immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab),
* Participant is found to be G6PD deficient
* Any drug listed in Table 2 in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug) and/or the Participant has a negative urine drug screen on retest by the pathology laboratory.
* Positive alcohol - breath test.

Specific to the study:

* Cardiac/QT risk:

  * A history of clinically significant ECG abnormalities
  * Known pre-existing prolongation of the QTc- interval considered clinically significant
  * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc-interval or any clinical condition known to prolong the QTcinterval. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
  * Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analysis.
* Known hypersensitivity to piperaquine or any of its excipients or 4-aminoquinolines, artemether or other artemisinin derivatives, lumefantrine, or other arylaminoalcohols.
* Unwillingness to abstain from consumption of quinine containing foods/beverages such as tonic water, lemon bitter, from inoculation (Day 0) to the end of the malaria treatment.
* Any history or presence of lactose intolerance.

On dosing days:

* Ingestion of any other drug, in the two weeks prior to dosing or during the blood sampling period that, in the opinion of the Medical Investigator, could compromise the study, e.g., through metabolic interactions, or analytical interference. However the Medical Investigator may permit the use of paracetamol for the treatment of headache or other pain. If drug therapy other than paracetamol or drug specified in the protocol, is required during the study periods, a decision to continue or discontinue the participant's participation will be made by the Medical Investigator, based on the nature of the medication and the time the medication was taken.
* Failure to conform to the requirements of the protocol.
* Detection of any drug listed in this protocol in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug).
* Vital signs outside the reference range and clinically significant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Prof, Principal Investigator — QIMR Berghofer Medical Research Institute
Locations (1):
- Q-Pharm Clinics, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collins KA, Wang CY, Adams M, Mitchell H, Rampton M, Elliott S, Reuling IJ, Bousema T, Sauerwein R, Chalon S, Mohrle JJ, McCarthy JS. A controlled human malaria infection model enabling evaluation of transmission-blocking interventions. J Clin Invest. 2018 Apr 2;128(4):1551-1562. doi: 10.1172/JCI98012. Epub 2018 Mar 12. PMID 29389671

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Piperaquine Phosphate After Infected Blood Malaria Challenge
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Piperaquine Phosphate After Infected Blood Malaria Challenge
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.03 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Successful Infection of Vector Mosquitoes Following Both Direct and Indirect Feeding on the Blood of Infected Participants
Description: Seven to ten days after blood feeding, mosquitoes will be dissected to check for oocysts in midgut preparations. For permanent preparations, oocysts will be stained with 0.1% mercurochrome in PBS for 5 to 60 mins then fixed in 1%glutaraldehyde or formaldehyde. Oocysts will be counted per mosquito dissected and recorded. Relationship between parasitemia, gametocytemia and mosquito infection (both oocyst prevalence and intensity) will be determined using generalized-linear mixed models. The number of mosquitoes dying prior to dissection will be recorded.
Time Frame: 7-10 days after blood feeding
Population: Transmission prevalence was too low to evaluate the ability of the drugs to inhibit mosquito-stage parasite development using direct skin-feeding assay (DFA), direct membrane-feeding assay (DMFA), or membrane feeding assay with serum replacement (MFA SR).
Arm/Group | Piperaquine Phosphate After Infected Blood Malaria Challenge
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety: Number of AEs
Description: Adverse events incidence
Time Frame: Blood stage Plasmodium falciparum Challenge Inoculum up to Day 31
Measure: Number; unit: Number of adverse events
Arm/Group | Piperaquine Phosphate After Infected Blood Malaria Challenge
Number analyzed (Participants) | 6
Number of adverse events | 40

ADVERSE EVENTS:
Time Frame: Overall study, up to Day 31
Arm/Group | Piperaquine Phosphate After Infected Blood Malaria Challenge
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Piperaquine Phosphate After Infected Blood Malaria Challenge (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hot flush (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Puncture site induration (Injury, poisoning and procedural complications) | 2 (3)
Puncture site reaction (Injury, poisoning and procedural complications) | 2 (3)
Lymphocyte count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (19)

LIMITATIONS AND CAVEATS:
The adult mosquito mortality was high and blood feeding rates were low in these experiments, indicating an unhealthy mosquito colony. Transmission data from this group were therefore excluded from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less